CLINICAL TRIAL: NCT00523432
Title: A Phase I Study of CCI-779 (Temsirolimus) in Combination With Topotecan in Patients With Gynecologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 15424A
Record Dates: First submitted 2007-08-29; First posted 2007-08-31 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Genital Neoplasms, Female
Keywords: ovarian cancer; cervical cancer; uterine cancer; fallopian tube cancer; endometrial cancer; vaginal cancer; peritoneal cancer; reproductive cancer
MeSH Terms: conditions — Genital Neoplasms, Female; Ovarian Neoplasms; Uterine Cervical Neoplasms; Uterine Neoplasms; Fallopian Tube Neoplasms; Endometrial Neoplasms; Vaginal Neoplasms | interventions — Topotecan; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Arm A will consist of subjects without prior pelvic radiation or with radiation to a field smaller than the whole pelvis. Subjects will receive weekly CCI-779 and topotecan at the assigned dose.
  Interventions: Drug: Topotecan; Drug: CCI-779 (temsirolimus)
- B (Experimental): Arm A will consist of subjects with prior whole pelvic radiation. Subjects will receive weekly CCI-779 and topotecan at the assigned dose.
  Interventions: Drug: Topotecan; Drug: CCI-779 (temsirolimus)

INTERVENTIONS:
Drug: Topotecan — Weekly doses via IV infusion. Dose will be assigned based on time of study entry.
Drug: CCI-779 (temsirolimus) — Weekly 25mg dose via IV infusion.

SUMMARY:
The aim of the trial is to determine the recommended phase II dose of weekly intravenous topotecan in combination with a fixed dose (25 mg or 15 mg) of weekly intravenous temsirolimus in patients with and without prior pelvic radiation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed recurrent or metastatic ovarian carcinoma, fallopian tube carcinoma, primary peritoneal carcinoma, cervical carcinoma, endometrial carcinoma, vulvar carcinoma, vaginal carcinoma, or carcinosarcoma of the ovary, endometrium or cervix.
* Prior Therapy: at least one and may have up to three prior cytotoxic chemotherapeutic regimens for the management of primary disease.
* Must be at least 18 years of age.
* GOG performance status must be 0 or 1.
* Patients must have adequate organ and marrow function as defined below:

  * hemoglobin ≥10g/dL
  * absolute neutrophil count ≥1,500/uL
  * platelets ≥100,000/uL
  * total bilirubin below the institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) below the institutional upper limit of normal
  * creatinine below the institutional upper limit of normal
  * cholesterol ≤ 350 mg/dL (fasting)
  * triglycerides ≤ 400 mg/dL (fasting)
  * albumin ≥ 3.0 mg/dL
* negative pregnancy test for women able to have children
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior therapy with topotecan
* More than 3 prior cytotoxic chemotherapeutic regimens or treatment with temsirolimus or any other mTOR inhibitor
* Concomitant hormonal therapy or radiation therapy
* Clinically significant infections or other medical problems of significant severity
* History of unstable angina or myocardial infarction within the past six months
* Known brain metastases unless the metastases have been controlled by prior surgery or radiotherapy, and the patient has been neurologically stable and off of steroids for at least 4 weeks.
* Any requirement for oxygen
* Cannot be receiving potent enzyme-inducing antiepileptic drugs (EIAEDs; e.g., phenytoin, carbamazepine, phenobarbital) nor any other potent CYP3A4 inducer such as rifampin or St. John's wort, as these may decrease temsirolimus levels. Use of agents that potently inhibit CYP3A4 (and hence may raise temsirolimus levels), such as ketoconazole, is discouraged, but not specifically prohibited.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-08; Primary Completion 2009-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Tolerability of regimen | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gini Fleming, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Result] Temkin SM, Yamada SD, Fleming GF. A phase I study of weekly temsirolimus and topotecan in the treatment of advanced and/or recurrent gynecologic malignancies. Gynecol Oncol. 2010 Jun;117(3):473-6. doi: 10.1016/j.ygyno.2010.02.022. Epub 2010 Mar 28. PMID 20347480
- [Derived] Yap TA, Carden CP, Kaye SB. Beyond chemotherapy: targeted therapies in ovarian cancer. Nat Rev Cancer. 2009 Mar;9(3):167-81. doi: 10.1038/nrc2583. PMID 19238149